CLINICAL TRIAL: NCT03820752
Title: Study of the Vaccination Coverage and Level of Protection Against Vaccine-preventable Infectious Diseases in Pediatric and Adult Risk Patients in a University Hospital
Brief Title: Vaccination Coverage and Level of Protection in Patients at Risk
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. dr. Corinne Vandermeulen, Principal Investigator, KU Leuven
Other Study IDs: UZVACC
Record Dates: First submitted 2014-12-01; First posted 2019-01-29 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Diabetes; Chronic Kidney Disease; Allergy; Cystic Fibrosis; Heart Disease
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Hypersensitivity; Cystic Fibrosis; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pediatric chronically ill patients: Through a questionnaire parents of chronically ill patients will be asked about the vaccination status of all recommended vaccines of their child. Also questions on disease, therapy and sociodemographic factors that can influence vaccination coverage will be asked.
  A blood sample to determine antibodies against measles, mumps, rubella and pertussis will be drawn from children who consent to sampling.
  The following groups of patients will be questioned: diabetes, allergy, congenital heart disease, cystic fibrosis, immunodeficiency and transplant patients, cancer patients.
- Adult chronically ill patients: Through a questionnaire chronically ill patients will be asked about their vaccination status of diphtheria, tetanus,pertussis, flu, pneumococcal and hepatitis B vaccine(s). Also questions on disease, therapy and sociodemographic factors that can influence vaccination coverage will be asked.
  A blood sample to determine antibodies against diphtheria, tetanus and pertussis will be drawn.
  The following groups of patients will be questioned: diabetes, chronic kidney disease, heart failure, COPD, immunodeficiency and transplant patients, HSCT patients.

SUMMARY:
The purpose of this study is to determine

1. vaccination coverage of recommended vaccines (routine childhood vaccines and vaccines against seasonal flu and pneumococci) in children with chronic diseases (allergy, cystic fibrosis, diabetes mellitus type 1, congenital heart disease, immunocompromised and solid organ transplant patients)
2. the level of protection against measles, mumps, rubella and pertussis in children with chronic diseases.
3. vaccination coverage of recommended vaccines (diphtheria, tetanus, pertussis and vaccines against seasonal flu and pneumococci) in adults with chronic diseases (nephropathy, diabetes mellitus, COPD, heart failure, HIV and solid organ transplant patients)
4. the level of protection against diphtheria, tetanus and pertussis in adults with chronic diseases.

DETAILED DESCRIPTION:
1. Chronically ill children

   1.1 What is the vaccination status for vaccines recommended by the Superior Health Council in pediatric chronically ill patients (2-16 years of age) who consult within the University hospital of Leuven?

   Patients with one of the following chronic conditions will be included:
   * Cystic fibrosis
   * Diabetes Mellitus type 1
   * Allergic constitution
   * Congenital heart disease
   * Solid-organ transplantpatients
   * Immunodeficiency (congenital or acquired)
   * Cancer

   The vaccination coverage for the following vaccines will be determined:
   * Poliomyelitis
   * Diphtheria
   * Tetanus
   * Pertussis
   * Haemophilus influenzae type b
   * Hepatitis B
   * Measles-Mumps-Rubella
   * Pneumococci
   * Meningococcal serogroup C
   * Rotavirus
   * Diphtheria-Tetanus-Polio: booster (older than 7 years)
   * Human papillomavirus (girls of 13 yrs)
   * Seasonal flu (cystic fibrosis, immunodeficiencies)

   Timeliness of the vaccines given will also be determined.

   1.2 Is the vaccination coverage of pediatric patients (2-16 years of age) comparable to the data on healthy children in 2012?

   1.3 What are possible factors that influence coverage in this specific patient populations?

   1.4 If the vaccination coverage is too low (below 90-95 percent), what are possbile solutions to increase the coverage rates within this group?

   1.5. Determine antibody titers in this same population for the following vaccine-preventable infectious diseases:
   * Measles
   * Mumps
   * Rubella
   * Pertussis

   1.6 Are antibody titers in this population similar to antibody titers measured in seroprevalence studies of healthy children in the same age group?
2. Adult patients at risk

2.1 What is the vaccinatiestatus for vaccines recommended by the Superior Health Council of adult patients at risk (over 18 years of age) who consult within the University hospital of Leuven?

Patients with one or more of the following chronic conditions will be included in the study:

* Chronic obstructive pulmonary disease (COPD)
* Heart failure
* Diabetes mellitus (Type 1 and 2)
* Chronic kidney disease (stadium IV and V)
* Solid organ Transplant patients
* HIV
* HSCT

The vaccination coverage for the following vaccines will be determined:

* Seasonal flu (yearly)
* Diphtheria-tetanus (date of last dose)
* Pneumococcus (1 dose/last dose before 5 years of age)
* Pertussis (1 dose)
* Hepatitis B (3 doses in specific risk groups)

2.2 Who immunizes these adult patients at risk?

2.3 What are possible risk factors who influences vaccination status in the adult population?

2.4 If the vaccination coverage is too low (below 90-95 percent), what are possible solutions to improve this coverage in these groups?

2.5 What are the antibody titers measured in the adult risk groups with a chronic condition for the following vaccine-preventable infectious diseases:

* Diphtheria
* Tetanus
* Pertussis

2.6 Are antibody titers measured in this population comparable to those of healthy subjects as measured in previous seroprevalence studies?

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients: be at least 2 years of age and maximum 16 ye
* adults patients: at least 18 years of age
* have a chronic condition

Exclusion Criteria:

-

Ages: 2 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronically ill patients (pediatric and adult) in follow-up at the University Hospital Leuven, Belgium
Sampling Method: Non-Probability Sample
Enrollment: 2179 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Proportion of pediatric chronically ill patients correctly vaccinated with the hexavalent (DTaP-IPV-Hib-HBV), pneumococcal, rotavirus, MMR and MenC vaccine according to the Belgian recommended vaccination schedule. | 5 years
  number of patients vaccinated compared to the entire group
Proportion of adult chronically ill patients correctly vaccinated diphtheria, tetanus, pneumococci, hepatitis B and influenza according to Belgian recommended vaccination schedule | 5 years
  number of patients vaccinated compared to the entire group

SECONDARY OUTCOMES:
Proportion of pediatric patients with antibodies against measles, mumps, rubella, diphtheria, tetanus and pertussis in children included in the study and who provided a blood sample | 5 years
  Determination of antibodies against measles, mumps, rubella and pertussis
Proportion of adult patients with antibodies against diphtheria, tetanus and pertussis. | 5 years
  Determination of antibodies against diphtheria, tetanus and pertussis

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Vandermeulen, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Result] Vandermeulen C, Roelants M, Theeten H, Depoorter AM, Van Damme P, Hoppenbrouwers K. Vaccination coverage in 14-year-old adolescents: documentation, timeliness, and sociodemographic determinants. Pediatrics. 2008 Mar;121(3):e428-34. doi: 10.1542/peds.2007-1415. PMID 18310163